CLINICAL TRIAL: NCT02743793
Title: A Prospective Cohort Study of Operationally Tolerant Allograft Recipients (ITN063ST)
Brief Title: A Cohort Study of Operationally Tolerant Allograft Recipients
Acronym: ALLTOL
Status: Terminated | Type: Observational
Why Stopped: COVID-19 pandemic and potential risks to study participants and study staff.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network); PPD Development, LP (Industry); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DAIT ITN063ST; UM1AI109565 (NIH)
Record Dates: First submitted 2016-04-06; First posted 2016-04-19 (Estimated); Results first posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-08

CONDITIONS: Kidney Transplant; Liver Transplant
Keywords: single organ liver or kidney allograft; operationally tolerant allograft recipients; longitudinal follow-up
MeSH Terms: interventions — Blood Specimen Collection; Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Operationally Tolerant Kidney or Liver Allograft Recipients: Operational tolerance at baseline is defined as:
  * An absence of any immunosuppressive therapy for ≥ 52 weeks prior to the screening visit;
  * No evidence of allograft rejection in the 52 weeks prior to the screening visit (Day 0), based on the participant's medical history; and
  * Normal and stable allograft function at screening visit defined as-
    * For liver transplant recipients: Liver function tests (ALT, GGT) both less than or equal to the upper limit of normal (ULN)
    * For kidney transplant recipients: Serum creatinine value corresponds to an estimated glomerular filtration rate (GFR) > 45 ml/min/1.73 m^2.
  Interventions: Procedure: Blood Draw

INTERVENTIONS:
Procedure: Blood Draw
  Other Names: Phlebotomy; Venesection; Venipuncture

SUMMARY:
Antirejection medicines, also known as immunosuppressive drugs, are prescribed to organ transplant recipients to prevent their bodies from rejecting the new organ. Some organ transplant recipients can stop taking anti-rejection medicines without rejecting their transplanted organ (this is called 'tolerance'). The purpose of this study will collect samples and data from 'tolerant' liver or kidney transplant recipients in order to find out:

The purpose of this study is to collect samples and data in order to find out:

* How long liver or kidney transplant recipients can remain tolerant;
* What happens in the tolerant recipient's body over time; and
* If there are patterns in the body that are linked to tolerance.

DETAILED DESCRIPTION:
This is a multi-center, prospective, observational study in which operationally tolerant recipients of liver or kidney allografts will be followed longitudinally, with annual collections of clinical data and biological samples. All participants will be followed for the duration of the study, regardless of changes in their tolerance status.

Participants will be recruited by three main pathways:

1. Tolerant participants from current and past Immune Tolerance Network (ITN) trials, including those who have already completed trial participation and those who are anticipated to complete trial participation,
2. Tolerant participants referred by ITN affiliated investigators, academic and community transplant physicians and directly through outreach to transplant affinity groups such as the National Kidney Foundation (NKF), and
3. Tolerant participants from the general transplant community who are reachable through general contact channels such as the ITN website, word-of-mouth referrals from existing participants, and social media.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of single organ liver or kidney allograft from a living or deceased donor;
* At screening, operationally tolerant, as defined by:

  * Absence of any immunosuppressive therapy for ≥52 weeks prior to the screening visit, and
  * No evidence of allograft rejection in the 52 weeks prior to the screening visit, based on the allograft recipient's medical history.
* Normal allograft function, defined as:

  * For liver transplant recipients: Liver function tests (ALT, GGT) both less than or equal to the upper limit of normal (ULN); and,
  * For kidney transplant recipients: Serum creatinine value corresponds to an estimated GFR > 45 ml/min/1.73 m^2.
* Receiving regular follow-up for a kidney or liver transplant by a local physician:

  --Participants must be willing to allow the study team to contact and share medical information with this local physician.
* Ability to sign informed consent.

Exclusion Criteria:

* Current malignancy requiring recent surgery, ongoing chemotherapy, or radiation;
* Transplant of another organ;
* Current drug or alcohol dependency;
* Any medical condition that in the opinion of the principal investigator would interfere with safe completion of the trial; and
* Inability to comply with the study visit schedule and required assessments.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Operationally tolerant recipients of liver or kidney allografts
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sindhu Chandran, M.D., Study Chair — Immune Tolerance Network (ITN)
Locations (5):
- United States (5):
  - University of California, San Francisco, San Francisco, California
  - Emory University School of Medicine, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Memorial Hospital of Chicago, Chicago, Illinois
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburg of UPMC, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data upon completion of the study in: Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: On average, within 24 months after database lock for the trial.
Access Criteria: Open access.
URL: https://www.immport.org/home

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Immune Tolerance Network (ITN) — https://www.immunetolerance.org/
- See also: ITN ALLTOL Study website — http://www.alltol.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 41 tolerant kidney and liver participants were recruited from June 2016 through February 2020 along three main pathways 1) from current and past Immune Tolerance Network (ITN) trials, 2) by ITN affiliation investigators, academic community transplant physicians, and through outreach to transplant affinity groups, and 3) from the general transplant community through media channels.
Pre-assignment Details: Informed consent was obtained from potentially eligible individuals who underwent a screening visit to determine eligibility.
Groups:
- Enrolled, Not Eligible: These participants were consented and enrolled into the study, but did not meet eligibility criteria.
- Accrued: These participations met all eligibility criteria and completed at least one mechanistic sample collection.
Period: Overall Study
Arm/Group | Enrolled, Not Eligible | Accrued
Started | 5 | 36
Completed | 0 | 0
Not Completed | 5 | 36
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Screen Failure | 4 | 0
Not completed — No Primary Care Physician | 0 | 1
Not completed — Travel/remote visits could not be performed at nursing facility | 0 | 1
Not completed — Study stopped due to COVID-19 pandemic | 0 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enrolled, Not Eligible | Accrued | Total
Number analyzed (Participants) | 5 | 36 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 9 | 11
  Between 18 and 65 years | 1 | 21 | 22
  >=65 years | 2 | 6 | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39 (29.4) | 40 (24.3) | 40 (24.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 20 | 20
  Male | 5 | 16 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 36 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 33 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 36 | 41
Duration of operational tolerance at time of enrollment. [Mean (Standard Deviation); unit: years] — To be considered for the trial, the participant had to have established operational tolerance. A participant is considered to have operational tolerance if they are off all immunosuppression medication while continuing to have stable allograft function and no rejection. For these participants, the date of operational tolerance is considered as 52 weeks from the participant's last documented dose of immunosuppression.
  years | 7.6 (5.07) | 8.1 (7.53) | 8.1 (7.32)
Alanine aminotransferase (ALT) [Mean (Standard Deviation); unit: U/L] — The ALT result from the screening visit. The measure is only relevant to liver recipients. The normal range is 7-41 U/L. Population: Number of participants analyzed based on number of participants with data available.
  U/L
    number analyzed (Participants) | 1 | 26 | 27
    (all) | 68.0 (NA) — Only one participant had an ALT result available. | 24.5 (11.98) | 26.1 (14.42)
Gamma glutamyltransferase (GGT) [Mean (Standard Deviation); unit: U/L] — The GGT result from the screening visit. The measure is only relevant to liver recipients. The normal range is 9-58 U/L. Population: Number of participants analyzed based on number of participants with data available.
  U/L
    number analyzed (Participants) | 1 | 25 | 26
    (all) | 18 (NA) — Only one participant had a GGT result available. | 32.4 (49.33) | 31.8 (48.42)
Creatinine [Mean (Standard Deviation); unit: mg/dL] — The creatinine result from the screening visit. The measure is only relevant to kidney recipients. The normal range for creatinine is 0.5-0.9 mg/dL for females and 0.6-1.2 mg/dL for males. Population: Number of participants analyzed based on number of participants with data available.
  mg/dL
    number analyzed (Participants) | 1 | 10 | 11
    (all) | 2.6 (NA) — Only one participant had a creatinine result available. | 1.3 (0.48) | 1.4 (0.60)

OUTCOME MEASURES:

1. Primary Outcome: Time to Loss of Operational Tolerance
Description: A participant is considered to have operational tolerance if they are off all immunosuppression medication while continuing to have stable allograft function and no rejection. For these participants, the date of operational tolerance is considered as 52 weeks from the participant's last documented dose of immunosuppression. A participant will be considered to have lost operational tolerance if they experience rejection, have loss of stable allograft function (in the absence of confounding factors), or restart immunosuppression. The endpoint was analyzed using Kaplan-Meier survival estimate and associated two-sided 95% confidence interval, using a delayed-entry model with left-truncation of survival times by censoring the time from achieving operational tolerance at the time of study enrollment. The survival estimate is at the time of the last of event.
Time Frame: From operational tolerance to ITN063ST study completion, assessed up to 60 months
Population: Participants who met all eligibility criteria and completed at least one mechanistic sample collection.
Measure: Mean (Standard Deviation); unit: Years to loss of operational tolerance
Groups:
- Accrued: These participants met all eligibility criteria and completed at least one mechanistic sample collection.
Arm/Group | Accrued
Number analyzed (Participants) | 36
Years to loss of operational tolerance | 6.6 (5.38)
Statistical Analysis 1: Comparison: Accrued; Test type: Other — No test was performed; Kaplan-Meier survival estimate = 64, 95% CI 2-sided [21.3 to 87.9] — Percent of participants that remained tolerant during study participation

2. Secondary Outcome: Time to Development of Anti-Human Leukocyte Antigen (HLA) Antibody or Donor Specific Antibodies (DSA)
Description: Time to development of either:
  * de novo HLA antibodies (anti-HLA Ab) post-transplant. Alloantibody is defined as an antibody produced following the introduction of an alloantigen into the system of an individual lacking that particular antigen; OR
  * Donor Specific Antibodies (DSA), a newly developed alloantibody that is against the donor organ.
  Alloantibodies are important mediators of acute and chronic rejection.
  **These data are not yet available.**
Time Frame: Day 0 (Study Enrollment) to Study Completion (Up to 3.7 years)
Reporting Status: Not Posted

3. Secondary Outcome: Number of Participants With Biopsy-Proven or Clinical Acute Rejection, Steroid Resistant Rejection and/or Chronic Rejection
Description: Number of participants with acute rejection, steroid resistant rejection and/or chronic rejection.
  Criteria employed for acute and chronic rejection: Banff guidelines.
Time Frame: Day 0 (Study Enrollment) to Study Completion (Up to 3.7 years)
Population: Participants who met all eligibility criteria and completed at least one mechanistic sample collection.
Measure: Count of Participants; unit: Participants
Arm/Group | Accrued
Number analyzed (Participants) | 36
Participants | 0

4. Secondary Outcome: Number of Participants With Graft Loss, Not Including Death With a Functioning Graft
Description: A participant is considered to have graft loss when the participant is retransplanted with another donor kidney, relisted for transplantation, or dies with a non-functioning graft.
Time Frame: Day 0 (Study Enrollment) to Study Completion (Up to 3.7 years)
Population: Participants who met all eligibility criteria and completed at least one mechanistic sample collection.
Measure: Count of Participants; unit: Participants
Arm/Group | Accrued
Number analyzed (Participants) | 36
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to 3.7 years.
Description: Only adverse events that met serious criteria were collected for this study.
  Inclusion: A serious adverse event (SAE) that occurred:
  * within 24 hours after a protocol-mandated blood draw, or
  * if an SAE occurred more than 24 hours after a protocol-mandated blood draw and was deemed as a possibly or definitely association with a protocol-mandated blood draw.
  Participants in the "Enrolled, Not Eligible" Arm/Group did not undergo any protocol mandated blood draws and are not represented.
Groups:
- Enrolled, Not Eligible: These participants were consented and enrolled into the study, but did not meet eligibility criteria. Only adverse events meeting serious criteria were collected for this study. A SAE is defined as "any adverse event that meets on or more serious criterion and occurs within 24 hours of the protocol mandated blood draw for research specimens. Those in the "Enrolled, Not Eligible" Arm/Group did not undergo any protocol mandated blood draws and so no adverse events will be reported for this Arm/Group.
- Accrued: Accrued participations met all eligibility criteria and completed at least one mechanistic sample collection. Only adverse events meeting serious criteria were collected for this study. An SAE is defined as "any adverse event that meets one or more serious criterion and occurs within 24 hours of the protocol mandated blood draw for research specimens".
Arm/Group | Enrolled, Not Eligible | Accrued
All-Cause Mortality (participants affected / at risk) | 1/5 | 1/36
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/36
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study team ended the study early due to the COVID-19 pandemic on March 24, 2020.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/93/NCT02743793/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-17): https://cdn.clinicaltrials.gov/large-docs/93/NCT02743793/SAP_001.pdf